CLINICAL TRIAL: NCT07289139
Title: PhEAR-Prehospital Emergency Airway Research.
Brief Title: Prehospital Emergency Airway Research.
Acronym: PhEAR
Status: Active, not recruiting | Type: Observational
Sponsor: Centro de Emergencias Sanitarias 061 Andalucía (Other)
Responsible Party: Principal Investigator, Cristina López López, MD Doctor of Medicine, Centro de Emergencias Sanitarias 061 Andalucía
Other Study IDs: 2025_CES_061_REG_PHEAR_V1
Record Dates: First submitted 2025-09-30; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Airway Management; Emergency
Keywords: airway management; critical care; emergency; endotracheal intubation
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The creation of an airway registry will allow an improvement in the quality of care, the safety of critically ill patients in pre-hospital situations, and a reduction in morbidity and mortality related to airway management.

DETAILED DESCRIPTION:
In the care of critically ill patients in prehospital emergency settings, advanced airway management (AAM) is essential to maintain airway patency and ensure adequate oxygenation and ventilation. In Andalusia, prehospital emergency teams are composed of a physician, a nurse, and an emergency medical technician (EMT), and they operate both ground units (advanced life support ambulances) and air units (medical helicopters).

AAM encompasses a wide range of processes, techniques, and complex decision-making interventions that can be key to favorable patient outcomes. However, if not performed correctly, these procedures can also lead to adverse events, poor prognosis, or preventable mortality.

The increasing complexity and technological sophistication of healthcare require health systems to improve and adapt in order to deliver safe, high-quality care, where continuity and an integrated vision of care are essential.

This comprehensive approach is made possible through the analysis of incidents recorded in registries, which play a key role in identifying failures in clinical practice and implementing new strategies to address them.

ELIGIBILITY:
Inclusion Criteria:

* All patients attended by the 061 Emergency Teams of Andalusia, with an "Assistance" type of request, who underwent any of the following techniques: manual ventilation, orotracheal intubation, supraglottic device insertion, or cricothyroidotomy

Exclusion Criteria:

* interhospital transfers,
* patients who recieve this techniques before de emergency team arrives

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients attended by the 061 Emergency Teams of Andalusia, with an "Assistance" type of request, who underwent any of the following techniques: manual ventilation, orotracheal intubation, supraglottic device insertion, or cricothyroidotomy
Sampling Method: Non-Probability Sample
Enrollment: 4300 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Calculate First-pass intubation success rate | 2 years
  Intubations performed on the first attempt divided by the total number of intubations

SECONDARY OUTCOMES:
Development and validation of an artificial intelligence-based predictive algorithm for prehospital difficult airway | 2 years
Identify early and late complications in patients undergoing prehospital advanced airway management | from admission until day 28 of hospitalization
  early complications (during out-of-hospital assistance), late complications (within the first 28 days after hospital admission)
calculate 28-day mortality | from admission until day 28 of hospitalization
  Number of patients with mortality within the first 28 days of hospital admission
hospital length of stay | one year
  number of days of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Emergencias Sanitarias 061 Andalucía, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No